CLINICAL TRIAL: NCT07176585
Title: A Prospective, Single-site, Single-group Value Study on the Diagnosis of Functional Myocardial Ischemia Based on IVUS Plaque Characteristics
Status: Completed | Type: Observational
Sponsor: Insight Lifetech Co., Ltd. (Industry)
Collaborators: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CIP-0201
Record Dates: First submitted 2025-09-01; First posted 2025-09-16 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Coronary Artery Disease
Keywords: IVUS; FFR; PCI; CAD
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to evaluate the accuracy of IVUS-calculated percent atheroma volume (PAV) for diagnosing functional myocardial ischemia, using FFR as the gold standard.

DETAILED DESCRIPTION:
This prospective, single-site, single-group target-value study aims to investigate the accuracy of intravascular ultrasound (IVUS)-based plaque characteristics in diagnosing functional myocardial ischemia, using coronary fractional flow reserve (FFR) as the gold standard.

ELIGIBILITY:
Inclusion Criteria:

1. Study participants must be at least 18 years of age and younger than 80 years of age, regardless of gender;
2. Stable coronary artery disease, unstable angina, or acute myocardial infarction (AMI ≥ 7 days);
3. Coronary angiography showed primary lesions with a visual stenosis of 30% to 90% in at least two coronary arteries ≥ 2.5 mm in diameter;
4. Willing to participate in the study and able to understand, read, and sign the informed consent form.

Exclusion Criteria:

1. STEMI as clinical presentation within 7 days;
2. Chronic Total Occlusion (CTO) as target vessel;
3. Significant contraindication to adenosine administration (e.g., atrioventricular block, severe asthma, etc.);
4. Study participants are currently participating in other drug or device clinical studies and have not achieved the study endpoints;
5. Pregnant or nursing;
6. Other situations considered by the investigator as unsuitable for participation in this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with multivessel coronary artery disease.
Sampling Method: Non-Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2025-09-23 (Actual); Primary Completion 2026-01-04 (Actual); Study Completion 2026-01-04 (Actual)

PRIMARY OUTCOMES:
Accuracy of PAV calculated from IVUS images on diagnosing functional myocardial ischemia | Intraoperative period（After coronary angiography, before the potential PCI）
  Using blood vessels as the research unit and FFR values measured by pressure microcatheters as a reference (FFR ≤ 0.80 is positive, FFR>0.8 is negative), evaluate the accuracy of PAV calculated from IVUS images on diagnosing functional myocardial ischemia PAV ≥ 39.0% is positive, PAV < 39.0% is negative).
Sensitivity and specificity of PAV calculated from IVUS images on diagnosing functional myocardial ischemia | Intraoperative period（After coronary angiography, before the potential PCI）
  Using blood vessels as the research unit and FFR values measured by pressure microcatheters as a reference (FFR ≤ 0.80 is positive, FFR>0.8 is negative), evaluate the sensitivity and specificity of PAV calculated from IVUS images on diagnosing functional myocardial ischemia (PAV ≥ 39.0% is positive, PAV < 39.0% is negative).

SECONDARY OUTCOMES:
The positive predictive value, negative predictive value, Receiver Operating Characteristic Curve (ROC) and Area Under the Curve (AUC) of PAV calculated from IVUS images on the diagnosis of functional myocardial ischemia. | Intraoperative period（After coronary angiography, before the potential PCI）
  Using blood vessels as the research unit and FFR values measured by pressure microcatheters as reference (FFR ≤ 0.80 is positive, FFR>0.8 is negative), evaluate the positive predictive value, negative predictive value, Receiver Operating Characteristic Curve (ROC), and Area Under the Curve (AUC) of PAV calculated from IVUS images on the diagnosis of functional myocardial ischemia (PAV ≥ 39.0% is positive, PAV < 39.0% is negative).
Accuracy, sensitivity, specificity, positive predictive value, and negative predictive value of Total Atheroma Volume (TAV) calculated from IVUS images on the diagnosis of functional myocardial ischemia | Intraoperative period（After coronary angiography, before the potential PCI）
  Using blood vessels as the research unit and FFR values measured by pressure microcatheters as a reference (FFR ≤ 0.80 is positive, FFR>0.8 is negative), evaluate the accuracy, sensitivity, specificity, positive predictive value, and negative predictive value of Total Atheroma Volume (TAV) calculated from IVUS images on the diagnosis of functional myocardial ischemia.
Accuracy, sensitivity, specificity, positive predictive value, and negative predictive value of Minimum Lumen Area (MLA) calculated from IVUS images on the diagnosis of functional myocardial ischemia | Intraoperative period（After coronary angiography, before the potential PCI）
  Using blood vessels as the research unit and FFR values measured by pressure microcatheters as a reference (FFR ≤ 0.80 is positive, FFR>0.8 is negative), evaluate the accuracy, sensitivity, specificity, positive predictive value, and negative predictive value of Minimum Lumen Area (MLA) calculated from IVUS images on the diagnosis of functional myocardial ischemia.
Accuracy, sensitivity, specificity, positive predictive value, and negative predictive value of Plaque Burden (PB) calculated from IVUS images on the diagnosis of functional myocardial ischemia | Intraoperative period（After coronary angiography, before the potential PCI）
  Using blood vessels as the research unit and FFR values measured by pressure microcatheters as a reference (FFR ≤ 0.80 is positive, FFR>0.8 is negative), evaluate the accuracy, sensitivity, specificity, positive predictive value, and negative predictive value of Plaque Burden (PB) calculated from IVUS images on the diagnosis of functional myocardial ischemia.
Accuracy, sensitivity, specificity, positive predictive value, and negative predictive value of Diameter Stenosis (DS%) calculated by Quantitative Coronary Angiography (QCA) on diagnosing functional myocardial ischemia | Intraoperative period（After coronary angiography, before the potential PCI）
  Using blood vessels as the research unit and FFR values measured by pressure microcatheters as a reference (FFR ≤ 0.80 is positive, FFR>0.8 is negative), evaluate the accuracy, sensitivity, specificity, positive predictive value, and negative predictive value of Diameter Stenosis degree (DS%) calculated by Quantitative Coronary Angiography (QCA) on diagnosing functional myocardial ischemia.
Correlation between PAV, TAV, MLA, PB, DS% and FFR in pairwise comparisons | Intraoperative period（After coronary angiography, before the potential PCI）
  Using blood vessels as the research unit, conducting Passing Bablok regression analysis and Pearson linear correlation analysis on Percent Atheroma Volume (PAV), Total Atheroma Volume (TAV), Minimum Lumen Area (MLA), Plaque Burden (PB), Diameter Stenosis degree (DS%) and Fractional Flow Reserve (FFR).
Correlation between PAV gradient calculated from IVUS images and FFR Pullback Pressure Gradient (PPG) | Intraoperative period（After coronary angiography, before the potential PCI）
  Using blood vessels as the research unit, PAV was calculated every 1mm along the vascular direction based on IVUS images, and FFR Pullback Pressure Gradient (PPG) distribution was calculated based on FFR pullback. The correlation between PAV gradient distribution along the vascular direction and FFR PPG was evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- Fuwai Hospital,Cams & Pumc, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided